CLINICAL TRIAL: NCT02068300
Title: 1,5-Anhydro-D-Glucitol Can Reflect Hypoglycemia in Patients With Well Controlled Type 2 Diabetes
Brief Title: The Role of 1.5-anhydro-D-glucitol as Clinical Biomarkers of Hypoglycemia in Patients With Diabetes
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hye Seung Jung, associate professor, Seoul National University Hospital
Other Study IDs: 1,5AG_Hypo
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes Mellitus With Hypoglycemia
Keywords: 1,5-anhydro-D-glucitol, hypoglycemia, surrogate marker
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood, urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the usefulness of plasma 1,5-anhydro-D-glucitol (1,5-AG) as a novel surrogate marker of hypoglycemia

DETAILED DESCRIPTION:
We enrolled well controlled diabetes patients who had hypoglycemic event at least one time more. All patients assess the risk of severe hypoglycemia and hypoglycemic unawareness using hypoglycemic awareness questionnaires (HYPO score). The patients who are treated with insulin agent were inserted sensor of continuous glucose monitoring systems under the skin during three days. We were analysed the correlation between 1,5-anhydro-D-glucitol and HYPO score.

ELIGIBILITY:
Inclusion Criteria:

* patients attending outpatients of department of endocrinology and metabolism, seoul national university hospital .(HbA1C <8%)
* The patients who treated with insulin or sulfonylureas at least 3month period
* In case fo sulfonylurea user, HbA1c was restricted under 8%
* The patients who had hypoglycemic event at least 3 months
* who has can be survey questionnaire
* who can insert continuous glucose monitoring system

Exclusion Criteria:

* renal dysfunction patients
* hepatic dysfunction patients
* who has any kind of diseases, operations, medical treatments that can affect glucose levels

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The correlation between 1,5-anhydro-D-glucitol and Modified Hypoglycemic score | within the least 3 months
  Modified hypoglycemic score was calculated by modified Clarke et al. questionnaire.

SECONDARY OUTCOMES:
The correlation between hypoglycemic percent of Continuous glucose monitoring system and modified hypoglycemic score in insulin using patients. | within at leat 3months
  Modified hypoglycemic score was calculated by modified Clarke et al. questionnaire.
  Continuous glucose monitoring system was performed to find hypoglycemic event and glycemic variability in insulin using patients.
The relation between glycemic variability indices such as MAGE of continuous glucose monitoring system and 1,5-AG in insulin using patients. | within at least 3months
  1,5-AG was measured from patient's serum. Continuous glucose monitoring system was performed to find hypoglycemic event and glycemic variability in insulin using patients.

OTHER OUTCOMES:
The plasma 1,5-anhydro-D-glucitol level may be a useful marker of daily glucose excursion in diabetes patients | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hye Seung Jung, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim MJ, Jung HS, Hwang-Bo Y, Cho SW, Jang HC, Kim SY, Park KS. Evaluation of 1,5-anhydroglucitol as a marker for glycemic variability in patients with type 2 diabetes mellitus. Acta Diabetol. 2013 Aug;50(4):505-10. doi: 10.1007/s00592-011-0302-0. Epub 2011 Jun 18. PMID 21688018